CLINICAL TRIAL: NCT03040258
Title: Interventions to Promote Healthy Eating and Physical Activity in Lebanese School Children Targeting Overweight and Obesity-Pilot Study
Brief Title: Interventions to Promote Healthy Eating and Physical Activity in Lebanese School Children Targeting Overweight and Obesity- Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NUT.NH.12
Record Dates: First submitted 2017-01-25; First posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Childhood Obesity
Keywords: School-based intervention
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group- Health-E-PALS-Pilot (Experimental): Group of students receiving the school-based intervention: Health-E-PALS (pilot), it consists of in class activities and lessons.
  Interventions: Other: Health-E-PALS-Pilot
- Control group (No Intervention): Group of students not receiving any intervention

INTERVENTIONS:
Other: Health-E-PALS-Pilot — Intervention to promote Healthy Eating and Physical Activity in Lebanese School-Children It comprises in class-activities, meetings with parents, improvement of school food service
  Arms: Intervention group- Health-E-PALS-Pilot

SUMMARY:
Evaluate the feasibility and effectiveness of a multi-component school-based intervention to promote healthy eating and physical activity with school children ages 9 to 11 years in Lebanon.

ELIGIBILITY:
Inclusion Criteria:

* Schoolchildren
* Aged 9 to 11 years

Exclusion Criteria:

- no exclusion criteria

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 374 (Actual)
Dates: Start 2008-03-10 (Actual); Primary Completion 2010-03-10 (Actual); Study Completion 2010-03-10 (Actual)

PRIMARY OUTCOMES:
Change in knowledge score | One school year
  Change in the knowledge scores (the sum of correct answers) based on a scored questionnaire delivered during pre- and -post assessment phases
Change in dietary habits | One school year
  Change in the percentage of children consuming sugary drinks, unhealthy and healthy snacks, fruits and vegetables/change in the percentage of children's physical activity frequency (self-reported in the questionnaires during pre- and -post assessment phases)
Change in self-efficacy score | One school year
  Change in the self-efficacy scores (the sum of correct answers) based on a scored questionnaire delivered during pre- and -post assessment phases

SECONDARY OUTCOMES:
Change in body weight status | One school year
  Change in Body Mass Index - BMI (in kg/m^2) at pre- and post-assesment.

CONTACTS AND LOCATIONS:
Overall Officials: Nahla Houalla, PhD, Principal Investigator — American University of Beirut Medical Center

IPD SHARING:
Plan to Share IPD: No